CLINICAL TRIAL: NCT05941117
Title: Effect of Weight Bearing Versus Non-weight Bearing Strengthening Exercises on Dynamic Balance in Knee Osteoarthritis Patients.
Brief Title: Effect of Exercises on Dynamic Balance in Knee Osteoarthritis Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Mahmoud Eldesoky, MSc, PhD candidate, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/003919
Record Dates: First submitted 2023-06-25; First posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Muscle Stretching Exercises; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- weight bearing exercises group (Active Comparator): 20 patients were assigned to this group with bilateral knees osteoarthritis, they received TENS, stretching exercises and weight bearing strengthening exercises.
  Interventions: Combination Product: stretching exercises; Combination Product: Transcutaneous electrical nerve stimulation; Combination Product: weight bearing strengthening exercises
- non-weight bearing exercises group (Active Comparator): 20 patients were assigned to this group with bilateral knees osteoarthritis, they received TENS, stretching exercises and Non-weight bearing strengthening exercises.
  Interventions: Combination Product: stretching exercises; Combination Product: Transcutaneous electrical nerve stimulation; Combination Product: Non-weight bearing strengthening exercises

INTERVENTIONS:
Combination Product: stretching exercises — stretching exercises for Hamstring, quadriceps and calf muscle for both lower limbs of the same patients. each exercise was repeated 5 times and each repetition hold for 30 seconds in the same session.
Combination Product: Transcutaneous electrical nerve stimulation — it is one of the electrical stimulation modalities which is used to relief pain, each patient receive it on both knees every session.
  Other Names: TENS
Combination Product: weight bearing strengthening exercises — strengthening exercises for quadriceps, gluteus maximus, gluteus Medius and calf muscle in the form of weight bearing from standing position each exercise was repeated for 10 times with 5 seconds hold in the same set and patient perform three sets in the same session for both lower limbs.
  Arms: weight bearing exercises group
Combination Product: Non-weight bearing strengthening exercises — strengthening exercises for quadriceps, gluteus maximus, gluteus Medius and calf muscle in the form of non-weight bearing from lying and setting positions each exercise was repeated for 10 times with 5 seconds hold in the same set and patient perform three sets in the same session for both lower limbs.
  Arms: non-weight bearing exercises group

SUMMARY:
This study is a randomized controlled trial which aims to compare the effect of weight bearing exercises and non-weight bearing exercises on the dynamic balance in knee osteoarthritis patients as 60 patients will divided in three groups where one group is control group and others two groups one of them perform weight bearing exercises and the other perform non weight bearing exercises.

ELIGIBILITY:
Inclusion Criteria:

* The patient's age > 50 years.
* Recent radiographs confirming the presence of knee OA, grade II-III (mild to moderate) Kellgren Lawrence (K/L).
* Body mass index (BMI) from 20 to 30 kg/m2.
* Met the American College of Rheumatology clinical criteria for mild to moderate knee OA.
* knee pain > 3 cm on a 10 cm visual analog scale (VAS) on most days of the previous week.
* Bilateral knee osteoarthritis.

Exclusion Criteria:

* Congenital or acquired inflammatory or neurological (systemic or local) diseases involving the knee.
* Patients who have mental or cognitive illness that interfere their ability to perform the exercises or the evaluation tests.
* Intra articular knee injection of steroids in the past 6 months.
* Patients who had received joint replacement surgery in either Knee or hip.
* Patients with rheumatoid arthritis.
* Patients who received physical therapy sessions on the knee in the past 6 months.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-10-25 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
change happened in the dynamic balance from the baseline | one day after the end of treatment
  Biodex Balance System which is a device used to measure the balance of a person who stand on the platform of the device that give a measurement called over all stability index where 0 score means the best balance and the largest number indicate bad balance.

SECONDARY OUTCOMES:
change happened in pain from the baseline | one day after the end of treatment
  Visual Analog Scale which is a scale for pain from 0 to 10 where 0 mean no pain and 10 is the maximum pain.
change happened in the joint angle repositioning from baseline | one day after the end of treatment
  Joint Repositioning Accuracy where the knee is moved passively to a certain angel and the patient hold it in this angle and then it moved to the start position and then the patient asked to move his knee joint actively to the previous the same previous angle then the absolute error between the true angle and the reproduced angle is measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No